CLINICAL TRIAL: NCT03094858
Title: Evaluation of a Smartphone Intervention to Reduce Sedentary Behavior
Acronym: SMARTpath
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The smartwatches we planned to use were discontinued.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7092
Record Dates: First submitted 2017-02-16; First posted 2017-03-29 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Risk Reduction Behavior
Keywords: Smartphone, sedentary behavior, smartphone intervention
MeSH Terms: conditions — Risk Reduction Behavior; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison group (Active Comparator): Equipment only comparison group will use Smartphone and Wristband to monitor sedentary behavior
  Interventions: Device: Wristband; Device: Smartphone
- Intervention group (Experimental): Intervention group will receive prompts from Smartphone to reduce sedentary behavior using information from Wristband
  Interventions: Device: Smartphone with prompts; Device: Wristband

INTERVENTIONS:
Device: Smartphone with prompts — Smartphone will be used to prompt randomly selected participants in intervention group to be active
  Other Names: Android Smartphone
  Arms: Intervention group
Device: Wristband — Wristband will monitor activity of all participants
  Other Names: Fitbit
Device: Smartphone — Smartphone will be used to monitor activity but prompts will not be given to randomly selected participants
  Other Names: Android
  Arms: Comparison group

SUMMARY:
Participants (N = 300) will be randomly assigned to: 1) an equipment-only comparison group that receives a smartphone and an activity monitor wristband but does not receive smartphone intervention prompts, or 2) the intervention group who will receive an activity monitor wristband that works in conjunction with a smartphone to reduce sedentary time via smartphone prompts during prolonged sedentary bouts. All participants will be provided with a Fitbit® wristband activity monitor and an Android smartphone on the same day of the week (i.e., Mondays). Participants will complete a 1-week baseline accelerometer and EMA period prior to the start of the intervention. Participants will be followed for 26 weeks after the intervention begins with follow-up visits at 6, 13, and 26 weeks. The primary outcome will be accelerometer-measured time spent in sedentary activity. Sedentary breaks, total active time, and time spent in light, moderate, and vigorous activity will be additionally evaluated as outcomes. Contextual variables and potential treatment mechanisms will be assessed via traditional questionnaire measurement and daily random EMAs at baseline and all follow-up visits. Brief smartphone-based daily diary assessments will be completed daily for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* A score of ≥ 4 on the REALM-SF85 indicating > 6th grade English literacy level, must be at least 18 years of age
* A BMI ≥ 25 (overweight/obese), not meeting current physical activity guidelines as measured by the 7-Day Physical Activity Recall
* Do not have a contraindication for physical activity based on the Physical Activity Readiness Questionnaire (PAR-Q)
* Able to attend all study visits, and possess a valid home address and a functioning telephone number.

Exclusion Criteria:

* Participants who have physical disabilities that restrict lower limb function and/or reading skills below a 7th grade reading level.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Accelerometer-measured sedentary time | One week
  Total accelerometer-measured time spent in sedentary activity

SECONDARY OUTCOMES:
Accelerometer-measured sedentary breaks | 26 weeks
  Accelerometer-measured time spent in sedentary activity
Accelerometer-measured total active time | 26 weeks
  Total active time
Accelerometer-measured time spent in light, moderate, and vigorous activity | 26 weeks
  Total time spent in light, moderate, and vigorous activity

CONTACTS AND LOCATIONS:
Overall Officials: Darla Kendzor, PhD, Principal Investigator — University of Oklahoma

IPD SHARING:
Plan to Share IPD: No